CLINICAL TRIAL: NCT04404764
Title: Characterization of the Clinical-epidemiological Profile of Patients With Spinal Muscular Atrophy (SMA) 5q Types II and III in Follow-up in the Brazilian Unified Public Health System: A Cross-sectional Observational Study (Registry)
Brief Title: Characterization of the Clinical-epidemiological Profile of Patients With SMA5q Types II and III: Observational Study
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Otavio Berwanger, Director, Hospital Israelita Albert Einstein
Other Study IDs: 27245419.0.0000.5259
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Spinal Muscular Atrophy type II; Spinal Muscular Atrophy type III; Mutation in SMN1; Nusinersen
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood | interventions — nusinersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treated with nusinersen at SUS: Patients with Spinal Muscular Atrophy (SMA) 5q types II and III treated with nusinersen in the Brazilian Unified Public Health System
  Interventions: Drug: Nusinersen Injectable Product
- With indication to receive nusinersen at SUS: Patients with Spinal Muscular Atrophy (SMA) 5q types II and III with indication, but not yet receiving nusinersen treatment in the Brazilian Unified Public Health System

INTERVENTIONS:
Drug: Nusinersen Injectable Product — The patient´s treatment is provided by SUS. The following dosage scheme of nurinersen is the one approved by ANVISA (Brazilian National Health Surveillance Agency): Nusinersen, 12 mg (5 mL) on days 0 (zero), 14 and 28. A fourth dose will be on day 63 with a maintenance dose once every 4 (four) months. The study will NOT have direct influence on the care received by patients. Data on adherence, interventions, hospitalizations, mechanical ventilation, procedures and adverse events will be obtained from the patients´ medical records.
  Other Names: Spinraza
  Groups: Treated with nusinersen at SUS

SUMMARY:
This study aims to characterize the clinical-epidemiological profile and baseline characteristics of patients with spinal muscular atrophy (SMA) 5q types II and III in follow-up at the Brazilian Unified Public Health System (SUS). The study data will be based on patients´ medical records from several Brazilian public hospitals, which will be defined by the Brazilian Ministry of Health (MS).

DETAILED DESCRIPTION:
This is a retrospective cross-sectional observational study to characterize the clinical and epidemiological profile of patients with spinal muscular atrophy (SMA) 5q types II and III, in follow-up at the Brazilian Unified Public Health System (SUS). This study aims to provide baseline data, which in the future may be used by the Brazilian Ministry of Health (MS) to assess the effectiveness of nusinersen. The clinical and epidemiological data will be collected from patients´ medical records, such as the score for the Hammersmith Functional Motor Scale - Expanded (HFMSE) and the Revised Upper Limb Module (RULM) at baseline, the WHO motor milestones at baseline, disease duration, age at the time of disease diagnosis, age at the time of disease screening, SMN2 (gene copy number), history of hospitalizations, history and characterization of previous surgical procedures, treatment dosage used, patient caregiver´s profile (ie, a family member or companion, who is responsible for taking care of the patient for most of the time). Other variables of interest that will also be collected are patient´s age and gender, geographic distribution, attending physician expertise and care structure where the patients were treated. The data acquisition will be performed using a paper and eletronic CRF (Case report Form). Written informed consent will be obtained from patients who meet the study elegibility criteria. The study will be performed in Brazilian public hospitals (centers) that are able to provide the treatment with nusinersen under the SUS scope. The total sample of patients and number of participating centers will be defined by the MS - SCTIE (Secretariat of Science, Technology and Strategic Supplies)/ DECIT (Department of Science and Technology). However, the initial estimation is a sample of 100 patients to be included in 10-15 centers.

ELIGIBILITY:
Patient Eligibility Criteria:

Inclusion Criteria:

* Participants of both sexes, in any age group, who have a clinical diagnosis of SMA 5q type II or type III, in follow-up at SUS, undergoing treatment with nusinersen or not
* Clinical and molecular diagnosis of SMA 5q type II (disease started after 6 months of age), or Clinical and molecular diagnosis of SMA 5q type III (disease started after 18 months of age)

Exclusion Criteria:

* Refusal to provide written informed consent (either the patient or a legal representative)
* Symptom onset after 19 years of age
* Need for invasive ventilatory support for 16 hours or more per day for more than 21 consecutive days
* Be participating or have participated in another clinical study aimed at specific treatment of SMA 5q other than with the drug nusinersen
* Having undergone treatment with gene therapy

Caretaker Eligibility Criteria:

Inclusion Criteria:

• First-degree family member or companion responsible for taking care of the patient with clinical diagnosis of SMA 5q type II or type III

Exclusion Criteria:

* Illiteracy
* Refusal to participate in the study

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Spinal Muscular Atrophy (SMA) 5q types II and III in follow-up in the Brazilian Unified Public Health System (SUS), undergoing treatment with nusinersen or not. For each patient included, a first-degree family member or companion responsible for taking care of the patient for most of the time will also be included, if they agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Expanded Hammersmith Functional Motor Scale | Baseline
  Hammersmith Functional Motor Scale-Expanded (HFMSE) scores range from 0 to 66, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Revised Upper Limb Module | In the inclusion of the study
  Revised Upper Limb Module (RULM) scores range from 0 to 37, with higher scores indicating better function.
WHO motor milestones | Unique evaluation at the time of inclusion
  The six World Health Organization (WHO) motor milestones are sitting without support, standing with assistance, hands and knees crawling, walking with assistance, standing alone, and walking alone.
Disease duration | At the time of inclusion in the study
  Time between diagnosis and age at inclusion in the study
Clinical features | Unique evaluation
  SMN2 (gene copy number);
History of hospitalizations | Documented in the period prior to the inclusion of the study
  Records of need for hospitalizations
History and characterization of previous surgical procedures | In the period prior to the inclusion of the study
  History of comorbidities
Treatment with nusinersen | Registration of the dose used at the time of inclusion in the study
  To undergo intrathecal administration of nusinersen at a dose of 12 mg

CONTACTS AND LOCATIONS:
Overall Officials: Otávio Berwanger, PhD, Study Director — Hospital Israelita Albert Einstein; Vanessa Teich, PhD, Study Chair — Hospital Israelita Albert Einstein; Edmar Zanoteli, PhD, Study Chair — University of Sao Paulo; Elice Batista, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (9):
- Brazil (9):
  - Universidade Federal de Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Hospital de Clínicas da Universidade Estadual de Campinas - Unicamp, Campinas
  - Associação Hospitalar de Prot Infancia Dr Raul Carneiro - Hospital Infantil Pequeno Príncipe, Curitiba
  - Hospital Infantil Dr. Albert Sabin, Fortaleza
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagão Gesteira da Universidade Federal do rio de Janeiro - UFRJ, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina de São Paulo - HCFMUSP, São Paulo
  - Universidade Federal de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No